CLINICAL TRIAL: NCT03868839
Title: An Open-label Feasibility Trial of Adjunctive Telmisartan in Patients With Treatment Resistant Schizophrenia
Brief Title: Telmisartan Pilot Study on Treatment Resistant Schizophrenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Xiaoduo Fan (Other)
Responsible Party: Sponsor-Investigator, Xiaoduo Fan, Associate Professor, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H00015574
Record Dates: First submitted 2019-03-06; First posted 2019-03-11 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia; Schizo Affective Disorder; Treatment-resistant Schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia, Treatment-Resistant | interventions — Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Telmisartan Pill (Experimental): Subjects will start telmisartan 40mg once a day during week 1; the dose will be increased to 80mg (target dose) or as tolerated during the remaining three weeks.
  Interventions: Drug: Telmisartan Pill

INTERVENTIONS:
Drug: Telmisartan Pill — telmisartan 40mg once a day during week 1; the dose will be increased to 80mg (target dose) or as tolerated during the remaining three weeks.
  Other Names: Micardis

SUMMARY:
This study is a 4-week pilot study for subjects with Schizophrenia or Schizoaffective Disorder who have not experienced a significant relief of symptoms from current anti-psychotic medication. The Investigators hypothesize that 4 weeks of telmisartan at 80mg daily will alter blood biomarkers for inflammation and oxidative stress after 4 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years inclusive.
* Primary diagnosis of Schizophrenia or Schizoaffective Disorder established by a structured psychiatric evaluation (MINI) based on Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-V) criteria.
* A Positive and Negative Syndrome Scale (PANSS) (Kay et al 1987) total score ≥ 70 with a score of > 4 on two or more of the following PANSS items: delusions, conceptual disorganization, hallucinatory behavior, suspiciousness, and unusual thought content.
* A score of ≥4 on the Clinical Global Impression-Severity (CGI-S) (Guy, 1976).
* Must have ongoing antipsychotic treatment for at least 8 weeks, with a stable dose for at least 4 weeks. Subjects who have failed to achieve clinically-recognized symptom reduction to at least 1 marketed antipsychotic agent at a therapeutic dose for ≥ 8 weeks during the past 12 months, will be eligible.
* Women of childbearing potential must have a negative pregnancy test performed at screening visit prior to receiving the study medication. Women enrolled in this trial must use single barrier contraception.

Exclusion Criteria:

* Psychiatrically unstable.
* Subjects with any clinically significant abnormalities as determined by medical history, physical exam, clinical and lab evaluation suggestive of an underlying disease state that may, in the opinion of the investigator, confound the results of study, increase risk to the subject, or lead to difficulty complying with the study plan.
* Current insulin treatment for diabetes.
* History of immunosuppression.
* Current or recent radiation or chemotherapy treatment for cancer.
* Chronic use of steroids (except local use or inhaler).
* Pregnancy or breastfeeding.
* Women who are planning to become pregnant.
* Use of diuretics, ACE inhibitors, spironolactone, potassium supplements, digoxin or warfarin because the possible drug-drug interaction with telmisartan.
* Tested positive for the urine drug screen.
* Subjects at imminent risk of suicide or injury to self or others, as per the opinion of the investigator, or history of significant suicide attempt within the last 6 months as per the Columbia Suicide Severity Rating Scale (C-SSRS).
* Subjects that have taken an investigational drug or taken part in a clinical trial within 30 days prior to screening.
* Subjects with a current (within the last 3 months) DSM-V diagnosis of alcohol or substance use disorder (excluding nicotine and caffeine) as established by the clinical assessment (MINI) at the screening visit will be excluded.
* Any other reason that, in the opinion of the investigator, would compromise patient safety or integrity of the study.
* Subjects with the lab values defined as exclusionary safety values.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoduo Fan, MD, MPH, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Psychotic Disorders Research Program, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telmisartan Pill
Started | 6
Completed | 5
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Study is terminated due to lack of funding.
Arm/Group | Telmisartan Pill
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.67 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4
  Black | 1
  Two or more races | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Changes in Blood Levels of Tumor Necrosis Factor Alpha
Description: Levels at week 4 minus levels at baseline
Time Frame: Baseline (week 0) to 4 weeks after initial dose
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Telmisartan Pill
Number analyzed (Participants) | 5
pg/mL | 1.10 (0.2377)

2. Primary Outcome: Changes in Blood Levels of Glutathione
Description: Levels at week 4 minus levels at baseline
Time Frame: Baseline (week 0) to 4 weeks after initial dose
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | Telmisartan Pill
Number analyzed (Participants) | 5
uM | 537.00 (196.404)

3. Primary Outcome: Changes in Blood Levels of Interleukin-6
Description: Levels at week 4 minus levels at baseline
Time Frame: Baseline (week 0) to 4 weeks after initial dose
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Telmisartan Pill
Number analyzed (Participants) | 5
pg/mL | 4.61 (3.4472)

4. Primary Outcome: Changes in Blood Levels of High Sensitivity C-Reactive Protein
Description: Levels at week 4 minus levels at baseline
Time Frame: Baseline (week 0) to 4 weeks after initial dose
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Telmisartan Pill
Number analyzed (Participants) | 5
mg/L | 2.34 (1.9642)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Telmisartan Pill
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telmisartan Pill (N=6)
Blurred vision (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The overall limitations and caveat is that this study is a pilot study with small sample size (6 subjects).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT03868839/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT03868839/SAP_001.pdf